CLINICAL TRIAL: NCT04125472
Title: Expanded Access Protocol to Provide Lumasiran to Patients With Primary Hyperoxaluria Type 1
Status: Approved for marketing | Type: Expanded Access
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-GO1-006
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Primary Hyperoxaluria
Keywords: Hyperoxaluria; Primary Hyperoxaluria; Kidney Diseases; Urologic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Metabolic Diseases; RNA Therapeutic; siRNA
MeSH Terms: conditions — Hyperoxaluria, Primary; Hyperoxaluria; Kidney Diseases; Urologic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Metabolic Diseases | interventions — lumasiran

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Lumasiran — Lumasiran administered as a subcutaneous (SC) injection
  Other Names: ALN-GO1

SUMMARY:
The purpose of this study is to provide expanded access to lumasiran for adults and pediatric patients with Primary Hyperoxaluria Type 1 (PH1),

DETAILED DESCRIPTION:
Choosing to participate in an expanded access program is an important personal decision. Talk with your doctor and family members or friends about deciding to join a research study. To learn more about this study, please have your doctor contact the study research staff using the Contacts provided. For general information, see the link provided in More Information.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Primary Hyperoxaluria Type 1

Exclusion Criteria:

* Clinically significant health concerns (with the exception of PH1)
* Received an investigational agent within 30 days before the first dose of lumasiran or are in follow-up of another clinical study
* Previously or currently participating in lumasiran clinical study
* History of liver transplant

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals

REFERENCES:
- See also: Information on the Early Access Program for Lumasiran — https://www.alnylam.com/medical-professional-resources/early-access-program/lumasiran/